CLINICAL TRIAL: NCT03151174
Title: Vitamin D, Strength, and Bone Density in Collegiate Athletes
Brief Title: Effects of Vitamin D Supplementation on Strength, Bone Density, and Injury Risk in Collegiate Athletes
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 17-009
Record Dates: First submitted 2017-05-01; First posted 2017-05-12 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Intervention Model Description: Subjects will either receive placebo, 5000IU, or 10000IU per day of Vitamin D for 8-12 weeks.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Any individuals involved in study measures will also be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Vitamin D - 10000IU (Experimental): These individuals have been categorized as Vitamin D deficient and will receive 10000IU of Vitamin D per day.
  Interventions: Drug: Vitamin D 10000 UNT
- Vitamin D - 5000IU (Experimental): These individuals have been categorized as Vitamin D insufficient and will receive 5000IU of Vitamin D per day.
  Interventions: Drug: Vitamin D 5000 UNT
- Placebo (No Intervention): These individuals have been categorized as Vitamin D sufficient and will receive placebo.

INTERVENTIONS:
Drug: Vitamin D 10000 UNT — 10000 IU Vitamin D per day
  Arms: Vitamin D - 10000IU
Drug: Vitamin D 5000 UNT — 5000 IU Vitamin D per day
  Arms: Vitamin D - 5000IU

SUMMARY:
The goal of this study is to determine whether Vitamin D supplementation improves strength and bone density, and reduces the risk of injury in collegiate athletes.

DETAILED DESCRIPTION:
Vitamin D is a hormone that is important for bone and muscle health. As such, not having enough vitamin D in your body is associated with increased risk of injury and reduced health and athletic performance. It is often recommended that individuals who have low levels of vitamin D take vitamin D supplements. However, the effects of vitamin D supplementation on health and strength gains in collegiate athletes are not known. The goal of this study is to determine whether vitamin D supplementation increases strength and bone density, while reducing the risk of injury in collegiate athletes. Fasting vitamin D concentrations will be measured and athletes will be supplemented daily with Vitamin D for 8-12 weeks. The amount of supplementation will depend on whether the athlete is categorized as sufficient (>30ng/ml), insufficient (20-35ng/ml), or deficient (<20ng/ml). Vitamin D concentrations, strength, bone density, and injury risk will be assessed before and after the intervention period.

ELIGIBILITY:
Inclusion Criteria:

* athlete for a sanctioned Virginia Tech sport

Exclusion Criteria:

* pregnant or trying to become pregnant, currently taking vitamin D (>600IU/day), calcium (>1000mg/dl), taking any performance enhancing supplements (example, creatine), or any other medication or nutritional supplements that might influence the study variables, cardiac or thyroid problems, have diabetes, or epilepsy

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2017-04-29 (Actual); Primary Completion 2018-05-15 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Strength | Up to 12 weeks
  Overall strength assessed via maximal strength testing. The specific tests may include the following, 1) one repetition max bench press (lbs) -, 2) one repetition max squat (lbs), 3) vertical jump test (feet), 4) broad jump test (feet), 5) dead lifts (lbs and repetition), 6) pull ups (repetition), 7) dips (repetition), and 8) shuttle time (test involving repeated sprints to and from marked points or lines - minutes/ seconds).

SECONDARY OUTCOMES:
Femur Bone Density | Up to 12 weeks
  Bone Density will be assessed in spine using Dual Energy X-ray Absorptiometry. T-scores will be determined.
Spine Bone Density | Up to 12 weeks
  Bone Density will be assessed in the hip (proximal femur) using Dual Energy X-ray Absorptiometry. T-scores will be determined.
Injury Occurence | Every week for up to 12 weeks
  New and current Injuries including bone breaks, muscle strains and sprains will be tracked via a questionnaire that will be filled out weekly. Subjects will report whether they had an injury, where the injury occurred on the body, the type of injury, as well as the date/ time of the injury and how the injury occurred.
  Number of injury

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Hulver, PhD, Principal Investigator — Virginia Polytechnic Institute and State University
Locations (1):
- Virginia Tech, Blacksburg, Virginia, United States

IPD SHARING:
Plan to Share IPD: No